CLINICAL TRIAL: NCT03273062
Title: A Double-blind, Placebo-controlled Clinical Trial to Evaluate the Effects of Catechol-O-Methyltransferase (COMT) Inhibition on Cognition and Neuropsychiatric Symptoms in Patients With a History of Acquired Brain Injuries
Brief Title: A Trial Evaluating Effects of COMT Inhibition in Patients With Acquired Brain Injury
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheppard Pratt Health System (Other)
Collaborators: Lieber Institute for Brain Development (Unknown)
Responsible Party: Principal Investigator, Robert Schloesser, MD, Executive Director, Sheppard Pratt-Lieber Research Institute, Inc., Sheppard Pratt Health System
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1087860-3
Record Dates: First submitted 2017-08-31; First posted 2017-09-06 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Brain Injuries; Brain Injuries, Traumatic; Brain Injury, Chronic
Keywords: Brain Injury; Traumatic Brain Injury; Acquired Brain Injury; Cognition; Neuropsychiatric Symptopms; COMT
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic; Brain Injury, Chronic | interventions — Tolcapone

STUDY DESIGN:
Intervention Model Description: Interventional clinical trial with a double-blind, randomized placebo-controlled crossover design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participant, respective care provider, as well as the investigator and research coordinator ("outcomes assessor") will all be blind to the order of placebo or medication (Tolcapone) administration in this two-arm, crossover study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Study Period 1 (Active Comparator): 15 days of Tolcapone 200mg TID
  OR
  Placebo Comparator 15 days of Placebo pill TID
  Interventions: Drug: Tolcapone 200 MG; Other: Placebo
- Study Period 2 (Placebo Comparator): 15 days of Placebo pill TID
  OR
  Active Comparator 15 days of Tolcapone 200mg TID
  Interventions: Drug: Tolcapone 200 MG; Other: Placebo

INTERVENTIONS:
Drug: Tolcapone 200 MG — Tolcapone 200 MG TID
  Other Names: Tasmar
Other: Placebo — Placebo, TID Placebo will be in capsules that are identical in appearance to intervention drug, Tolcapone.

SUMMARY:
This is a follow-up study for an ongoing open label trial conducted by the Sheppard Pratt-Lieber Research Institute utilizing the catechol-O-methyl-transferase (COMT) inhibitor Tolcapone to evaluate its effects on cognition and neuropsychiatric symptoms in patients with brain injuries (BI).

In this study, investigators will conduct a double-blind, placebo-controlled clinical trial utilizing a crossover design to study the effects of two weeks of Tolcapone 200mg administered three times a day (total of 600mg/day) on cognitive performance. Physical, emotional, cognitive and social functioning will also be evaluated through participant and proxy report. The investigators are planning to randomize a total of 12 patients with a history of acquired brain injury (BI).

DETAILED DESCRIPTION:
The proposed study is a follow-up study for an ongoing open label trial conducted by the Sheppard Pratt-Lieber Research Institute utilizing the catechol-O-methyl-transferase (COMT) inhibitor Tolcapone to evaluate its effects on cognition and neuropsychiatric symptoms in patients with brain injuries (BI).

The outcome measures utilized in this study were chosen based on the available data from the currently ongoing open-label clinical trial. The proposed study will utilize the same study medication at the same dose and frequency. In addition, the length of administration of study medication (two weeks) is identical. In the proposed study, investigators will conduct a double-blind, placebo-controlled clinical trial utilizing a crossover design to study the effects of two weeks of Tolcapone 200mg administered three times a day (total of 600mg/day) on cognitive performance. Physical, emotional, cognitive and social functioning will be evaluated through participant and proxy report. The investigators are planning to randomize a total of 12 patients with BI.

The cross-over design requires two 2-week long study periods during which the participant receives either Tolcapone two 100mg capsules three times a day (total of 600mg/day) or placebo. Participants will be randomly assigned to two sequence groups either starting with Tolcapone treatment (T-P group) or placebo (P-T group). Investigators and participants will be blind to the study group assignment and hence blind to the treatment (Tolcapone vs. placebo) that subjects receive at a given time. The study periods are separated by a "washout period" that is at least two weeks and maximally 4 weeks long to reduce the potential for carryover effects. Patient reported outcomes will be obtained a total of four times, twice prior to the start of each respective study period (Pre-Study Period Visits I & II) as well as at the end of each study period (Outcome Measures Visits I & II). Cognitive outcome measures will be obtained twice throughout the study, at the end of each respective study period (Outcome Measures Visits I & II).

ELIGIBILITY:
Inclusion Criteria:

* Capacity for written informed consent
* Ages 18-70 years, inclusive
* Diagnosis of a BI including mild, moderate, or severe TBI, or other acquired BI and post-BI development of neuropsychiatric complaints.
* Index event resulting in Traumatic or Acquired Brain Injury occurred >12 months prior to trial initiation
* A current or former patient at the clinics of the Sheppard Pratt Neuropsychiatry Program or another Sheppard Pratt outpatient clinic with medical documentation of BI
* Proficient in the English language
* Available to come to Sheppard Pratt Towson for the baseline evaluation and testing and for the duration of the protocol
* Stable neurological and psychiatric symptomatology for two months prior to trial initiation as determined by the referring Sheppard Pratt physician.
* Stable medication dose and regimen for two months prior to trial initiation (based on a review of medical chart)

Exclusion Criteria:

* History of, or active, liver disease or abnormal liver function tests-if the patient currently has elevated Alanine Transaminase (ALT) or Aspartate Transaminase (AST) levels that exceed 2 times the upper limit of normal [Normal Reference Ranges ALT (Male: 4-40 IU/L, Female: 4-40 IU/L), AST (Male: 4-31 IU/L, Female: 4-37 IU/L) or the ratio of AST: ALT has exceeded 2:1
* Uncontrolled hypo-or hypertension based on Joint National Committee criteria (JNC7) Hypotension: Systolic <90mmHg or diastolic <60mmHg Hypertension: Systolic >140mmHg or diastolic >90 mmHg)
* Active alcohol use disorder, as defined by DSM-5, of any severity mild, moderate, or severe
* Active illicit substance use, resulting in a substance use disorder as defined by DSM-5, of any severity mild, moderate, or severe
* Patient is currently taking Tolcapone or any of the following medications that can interact with Tolcapone resulting in an adverse event: another COMT inhibitor, benserazide, α-methyldopa, Dobutamine, Apomorphine, Isoproterenol, Clozapine, MAO inhibitor
* Known allergy or serious adverse reaction to Tolcapone
* Participated in any investigational drug trial within the past 30 days.
* Pregnant or planning to become pregnant during the study period
* Breastfeeding or planning to breastfeed during the study period.
* Presence of severe pre-morbid/pre-BI cognitive impairment or behavioral dysfunction, as per informant or medical documentation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2017-07-20 (Actual); Primary Completion 2018-07-20 (Estimated); Study Completion 2018-07-20 (Estimated)

PRIMARY OUTCOMES:
NIH Toolbox Fluid Cognitive Battery | Administered on the 14th day of Tolcapone or Placebo treatment (i.e. during each Outcome Measures Visit).
  This battery is a measure of cognitive performance derived from a battery of five cognitive assessments.

SECONDARY OUTCOMES:
TBI Quality-of-Life Measurement System | Administered prior to the start of Tolcapone oe Placebo treatment (i.e. during each Pre-Study Visit) and on the 14th day of Tolcapone or Placebo treatment (i.e. during each Outcome Measures Visit).
  A patient reported outcome measure assessing physical, emotional, cognitive and social functioning. Quality of Life Measure is a computer adaptive questionnaire.
Frontal Systems Behavior Scale | Administered prior to the start of Tolcapone oe Placebo treatment (i.e. during each Pre-Study Visit) and on the 14th day of Tolcapone or Placebo treatment (i.e. during each Outcome Measures Visit).
  A patient reported outcome measure, and proxy reported outcome measure, assessing neuropsychiatric symptoms associated with prefrontal cortical dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Schloesser, MD, Principal Investigator — Sheppard Pratt Health System
Locations (1):
- Sheppard Pratt Health System, Towson, Maryland, United States

IPD SHARING:
Plan to Share IPD: No